CLINICAL TRIAL: NCT07074873
Title: Assessment of Pelvic Floor Muscle Activation in Adolescents With Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024 - 1550
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Floor Muscle Activation; Idiopathic Scoliosis
Keywords: Pelvic Floor Muscle Activation; Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with adolescent idiopathic scoliosis: Patients aged 10-18 years diagnosed with adolescent idiopathic scoliosis (Participants who have undergone X-rays for screening purposes (family history of scoliosis, postural abnormalities in appearance) at Istanbul Gaziosmanpaşa Training and Research Hospital and whose Cobb angles are above 10 degrees and will be included.)
  Interventions: Other: Descriptive information form; Other: Health-Related Quality of Life Assessment; Diagnostic Test: Trunk rotation angle; Diagnostic Test: Cobb angle measurement; Diagnostic Test: Pelvic floor muscle activation measurement
- Healthy participants aged 10-18 with Cobb angle of less than 10 degrees: Participants who have undergone X-rays for screening purposes (family history of scoliosis, postural abnormalities in appearance) at Istanbul Gaziosmanpaşa Training and Research Hospital and whose Cobb angles are below 10 degrees will be included.
  Interventions: Other: Descriptive information form; Other: Health-Related Quality of Life Assessment; Diagnostic Test: Trunk rotation angle; Diagnostic Test: Cobb angle measurement; Diagnostic Test: Pelvic floor muscle activation measurement

INTERVENTIONS:
Other: Descriptive information form — The age, gender, height, weight, body mass index, age at menarche, time of initial diagnosis, how it was detected (medical history), family history (genealogy), dominant hand use, exercise habits (type of sport and duration), and corset use of individuals participating in the study will be recorded.
  Other Names: Assessment Tool
Other: Health-Related Quality of Life Assessment — The Paediatric Quality of Life Inventory is a valid and reliable health-related quality of life questionnaire used for children. This inventory, which has been adapted into Turkish, consists of two forms for children and families. Both forms include sections on physical functioning (8 items), emotional functioning (5 items), social functioning (5 items), and school functioning (5 items). Scoring is done on a scale of 0-5 for each question (0 = Never causes a problem, 1 = Rarely causes a problem, 2 = Sometimes causes a problem, 3 = Often causes a problem, and 4 = Always causes a problem). The total score of the inventory ranges from 0 to 100 points (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0). A high score indicates better health-related quality of life. Since our study population is aged 10-18, the inventories developed for the 8-12 and 13-18 age groups will be used.
  Other Names: Paediatric Quality of Life Inventory
Diagnostic Test: Trunk rotation angle — The Adam's Forward Bend Test is used as the primary assessment test in the clinical examination of scoliosis patients. In our study, the scoliometer assessment will be performed on the study group while the subjects are standing with equal weight on both feet. Patients will be asked to bend forward so that their shoulder level is aligned with their hip level (body parallel to the ground), and measurements will be taken with the scoliometer, with the highest degree recorded. The Baseline Scoliometer will be used for evaluations.
Diagnostic Test: Cobb angle measurement — The Cobb angle allows for the evaluation of deformity in the frontal plane in scoliosis. It is obtained by measuring the lateral flexion angle of scoliosis from a standing spinal X-ray taken in the posterior-anterior direction. The angle between the perpendicular lines connecting the parallel line drawn from the upper edge of the uppermost vertebra (upper vertebra) involved in the curvature and the parallel line drawn from the lower edge of the lowest vertebra (lower vertebra) gives the Cobb angle. In our study, the Cobb angle will be recorded from the spinal X-ray.
  Other Names: Cobb method
Diagnostic Test: Pelvic floor muscle activation measurement — The physiotherapist will position the child in a supine position with the knees flexed at 140 degrees, the soles of the feet in contact with the bed, and the thighs and feet approximately 30 centimetres apart. Two surface electrodes will be placed at the 3 and 7 o'clock positions on the perineal region, and a 30×30 mm single-use electrode will be placed on the right thigh as a reference electrode. Children will be taught to contract the correct pelvic floor muscles to move in the ventral and cranial directions. The 'Work-Rest Assessment,' lasting a total of 55 seconds, will be applied to each child using the same device. First, children will be asked to relax their pelvic floor muscles. Then, 5 seconds of contraction (work) and 5 seconds of relaxation (rest) will be performed, and a total of 10 cycles of contraction and relaxation of the pelvic floor muscles will be requested. The device provides a report of the data in graphical and numerical form at the end of the measurement.

SUMMARY:
Adolescent idiopathic scoliosis is a three-dimensional deformity of the spine with a curvature of at least 10° on radiography, accompanied by rotation, seen in children aged 10-18 years, the cause of which is unknown. The pelvic floor consists of muscles and connective tissue in the shape of an equilateral triangle bounded by the symphysis pubis at the front, the sacrum at the back, and the ischial spines at the sides. The pelvic floor supports the pelvic organs, controls intra-abdominal pressure, maintains urinary and faecal control, and provides dynamic support to the body in conjunction with other core muscles. The aim of our study is to investigate pelvic floor muscle activation in adolescents with idiopathic scoliosis. Our study will include volunteers diagnosed with adolescent idiopathic scoliosis at Istanbul Gaziosmanpaşa Training and Research Hospital who have been referred to the Spine Unit of Gaziosmanpaşa Physical Therapy Training and Research Hospital for control purposes (presence of scoliosis in the family, postural abnormalities in appearance). X-rays will be taken, and volunteers with Cobb angles below 10 degrees will be included. Taking into account a 15% loss of the calculated sample, a total of 19 patients will be included in the study. The study group will consist of individuals diagnosed with adolescent idiopathic scoliosis, and the control group will consist of healthy individuals without spinal deformities. Each individual who agrees to participate in the study will undergo evaluations. For the study group, evaluations will include Cobb angle (radiography), trunk rotation angle (forward bending test), pelvic floor muscle activation (Neurotrac Myoplus 4 Pro) for both groups, and health-related quality of life (Paediatric Quality of Life Inventory).

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis is a three-dimensional deformity of the spine with a curvature of at least 10° on radiography, accompanied by rotation, seen in children aged 10-18 years, the cause of which is unknown. The pelvic floor consists of muscles and connective tissue in the shape of an equilateral triangle bounded by the symphysis pubis at the front, the sacrum at the back, and the ischial spines at the sides. The pelvic floor supports the pelvic organs, controls intra-abdominal pressure, maintains urinary and faecal control, and provides dynamic support to the body in conjunction with other core muscles. The aim of our study is to investigate pelvic floor muscle activation in adolescents with idiopathic scoliosis.

Our study will include volunteers diagnosed with adolescent idiopathic scoliosis at Istanbul Gaziosmanpaşa Training and Research Hospital who have been referred to the Spine Unit of Gaziosmanpaşa Physical Therapy Training and Research Hospital for control purposes (presence of scoliosis in the family, postural abnormalities in appearance). X-rays will be taken, and volunteers with Cobb angles below 10 degrees will be included. Taking into account a 15% loss of the calculated sample, a total of 19 patients will be included in the study. The study group will consist of individuals diagnosed with adolescent idiopathic scoliosis, and the control group will consist of healthy individuals without spinal deformities. Each individual who agrees to participate in the study will undergo evaluations. For the study group, evaluations will include Cobb angle (radiography), trunk rotation angle (forward bending test), pelvic floor muscle activation (Neurotrac Myoplus 4 Pro) for both groups, and health-related quality of life (Paediatric Quality of Life Inventory).

Descriptive information form: The age, gender, height, weight, body mass index, age at menarche, time of initial diagnosis, how it was detected (medical history), family history (genealogy), dominant hand use, exercise habits (type of sport and duration), and corset use of individuals participating in the study will be recorded.

Health-Related Quality of Life Assessment: The Paediatric Quality of Life Inventory is a valid and reliable health-related quality of life questionnaire used for children. This inventory, which has been adapted into Turkish, consists of two forms for children and families. Both forms include sections on physical functioning (8 items), emotional functioning (5 items), social functioning (5 items), and school functioning (5 items). Scoring is done on a scale of 0-5 for each question (0 = Never causes a problem, 1 = Rarely causes a problem, 2 = Sometimes causes a problem, 3 = Often causes a problem, and 4 = Always causes a problem). The total score of the inventory ranges from 0 to 100 points (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0). A high score indicates better health-related quality of life. Since our study population is aged 10-18, the inventories developed for the 8-12 and 13-18 age groups will be used.

Trunk rotation angle: The Adam's Forward Bend Test is used as the primary assessment test in the clinical examination of scoliosis patients. In our study, the scoliometer assessment will be performed on the study group while the subjects are standing with equal weight on both feet. Patients will be asked to bend forward so that their shoulder level is aligned with their hip level (body parallel to the ground), and measurements will be taken with the scoliometer, with the highest degree recorded. The Baseline Scoliometer will be used for evaluations.

Cobb angle measurement: The Cobb angle allows for the evaluation of deformity in the frontal plane in scoliosis. It is obtained by measuring the lateral flexion angle of scoliosis from a standing spinal X-ray taken in the posterior-anterior direction. The angle between the perpendicular lines connecting the parallel line drawn from the upper edge of the uppermost vertebra (upper vertebra) involved in the curvature and the parallel line drawn from the lower edge of the lowest vertebra (lower vertebra) gives the Cobb angle . In our study, the Cobb angle will be recorded from the spinal X-ray.

Pelvic floor muscle activation measurement: Electromyographic measurement is the best-known non-invasive and practical method for measuring pelvic floor muscle activity (6). In our study, children's pelvic floor muscle activations will be assessed by a physiotherapist using the NeuroTrac Myoplus Pro4 device. The measurement will be performed in a room where no one else is present except the child and their parent. At the beginning, parents and the child will be informed about how the measurement will be performed. Before the measurement is taken, the child will be asked to completely empty their bladder. The physiotherapist will position the child in a supine position with the knees flexed at 140 degrees, the soles of the feet in contact with the bed, and the thighs and feet approximately 30 centimetres apart. Two surface electrodes will be placed at the 3 and 7 o'clock positions on the perineal region, and a 30×30 mm single-use electrode will be placed on the right thigh as a reference electrode. Children will be taught to contract the correct pelvic floor muscles to move in the ventral and cranial directions. The 'Work-Rest Assessment,' lasting a total of 55 seconds, will be applied to each child using the same device. First, children will be asked to relax their pelvic floor muscles. Then, 5 seconds of contraction (work) and 5 seconds of relaxation (rest) will be performed, and a total of 10 cycles of contraction and relaxation of the pelvic floor muscles will be requested. The device provides a report of the data in graphical and numerical form at the end of the measurement.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 10-18 diagnosed with adolescent idiopathic scoliosis (Study Group)
* Adolescents aged 10-18 not diagnosed with adolescent idiopathic scoliosis (Healthy partcipants) (Control Group)
* No neurological or psychiatric disorders (Study and Control Group)
* Parents and children must volunteer to participate in the study (Study and Control Group)

Exclusion Criteria: For both Study and Control Group

* Having undergone surgery on the chest, abdomen or pelvic area
* Having undergone scoliosis surgery or being a candidate for surgery
* Having any mental health issues
* Having scoliosis that is not idiopathic but has arisen for other reasons (neurological, congenital, etc.)
* Having a diagnosis of urinary incontinence
* Being actively involved in sports

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Our study will include volunteers who have been diagnosed with adolescent idiopathic scoliosis at Istanbul Gaziosmanpaşa Training and Research Hospital and referred to the Spine Unit at Gaziosmanpaşa Physical Therapy Training and Research Hospital. Participants who volunteer to participate in the study will be selected based on the following inclusion and exclusion criteria.
  The control group of our study will include volunteers who underwent X-ray examinations for control purposes (presence of scoliosis in the family, postural abnormalities in appearance) at Istanbul Gaziosmanpaşa Training and Research Hospital and whose Cobb angles were below 10 degrees.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle activation measurement | Within one month of receiving a diagnosis and agreeing to volunteer
  Electromyographic measurement is the best-known non-invasive and practical method for measuring pelvic floor muscle activity. In our study, children's pelvic floor muscle activations will be assessed by a physiotherapist using the NeuroTrac Myoplus Pro4 device. Two surface electrodes will be placed at the 3 and 7 o'clock positions on the perineal region, and a 30×30 mm single-use electrode will be placed on the right thigh as a reference electrode. Children will be taught to contract the correct pelvic floor muscles to move in the ventral and cranial directions. The 'Work-Rest Assessment,' lasting a total of 55 seconds, will be applied to each child using the same device. First, children will be asked to relax their pelvic floor muscles. Then, 5 seconds of contraction (work) and 5 seconds of relaxation (rest) will be performed, and a total of 10 cycles of contraction and relaxation of the pelvic floor muscles will be requested. The device provides a report of the data in graphical.

SECONDARY OUTCOMES:
Health-Related Quality of Life Assessment | Within one month of receiving a diagnosis and agreeing to volunteer
  The Paediatric Quality of Life Inventory is a valid and reliable health-related quality of life questionnaire used for children. This inventory, which has been adapted into Turkish, consists of two forms for children and families. Both forms include sections on physical functioning (8 items), emotional functioning (5 items), social functioning (5 items), and school functioning (5 items). Scoring is done on a scale of 0-5 for each question (0 = Never causes a problem, 1 = Rarely causes a problem, 2 = Sometimes causes a problem, 3 = Often causes a problem, and 4 = Always causes a problem). The total score of the inventory ranges from 0 to 100 points (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0). A high score indicates better health-related quality of life (2). Since our study population is aged 10-18, the inventories developed for the 8-12 and 13-18 age groups will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, Gaziosmanpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hodges PW, Sapsford R, Pengel LH. Postural and respiratory functions of the pelvic floor muscles. Neurourol Urodyn. 2007;26(3):362-71. doi: 10.1002/nau.20232. PMID 17304528
- [Background] Sapsford R. Rehabilitation of pelvic floor muscles utilizing trunk stabilization. Man Ther. 2004 Feb;9(1):3-12. doi: 10.1016/s1356-689x(03)00131-0. PMID 14723856
- [Background] Koenig I, Luginbuehl H, Radlinger L. Reliability of pelvic floor muscle electromyography tested on healthy women and women with pelvic floor muscle dysfunction. Ann Phys Rehabil Med. 2017 Nov;60(6):382-386. doi: 10.1016/j.rehab.2017.04.002. Epub 2017 Jul 14. PMID 28716538